CLINICAL TRIAL: NCT04408196
Title: Effects of Social Distancing on the Quality of Life and on the Emotional-affective Sphere of Caregivers and Patients Hospitalized in Residential Rehabilitation Departments: an Observational Study.
Brief Title: QoL and the Emotional-affective Sphere in Rehabilitation Setting During COVID-19 Quarantine
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, Md, PhD, Principal Investigator, Head of Rehabilitation Unit, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG_socialdistancing_COVID-19
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Rehabilitation
Keywords: rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 100 patients admitted to an inpatient rehabilitation facility
- Caregivers: 100 caregivers of patients admitted to an inpatient rehabilitation facility

SUMMARY:
Coronavirus disease (COVID-19) is caused by the Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) virus. This virus was identified in December 2019 in the Chinese city of Wuhan, in the province of Hubei, where it determined a state of health emergency proclaimed by China on January 30, 2020.

Since February 2020, Italy has been involved in the emergency of the COVID-19 infection, with devastating consequences for the health of the population and the economy of our country. As published by the Italian National Institute of Health, the starting date of the symptoms dates back to the end of January, the first case diagnosed dates back to 21 February 2020 while the first cases of home isolation date back to March 1st, 2020. On March 30, 2020, there were 101739 positive subjects and 11591 deaths (Civil Protection data).

According to data published by the World Health Organization, most people with COVID-19 develop a flu-like form, 14% develop a severe form that requires hospitalization and oxygen therapy and 5% require an ICU admission.

The emergency from Covid19 made it necessary to provide institutional social distancing conditions which resulted in rehabilitation departments being prohibited from visiting patients by family members and/or caregivers. This event, although necessary, led to the first moment of discomfort on the part of patients and family members; to overcome this reaction "technological" solutions were found, trying to give continuity to the contact between the patient and the family member through the use of video calls. Despite this, the COVID-19 emergency and the limitations resulting from social distancing likely have an impact on both patients and family members/caregivers that needs to be assessed.

DETAILED DESCRIPTION:
Aims:

The study aims to measure the quality of life (QoL) and the emotional-affective sphere of patients, currently hospitalized in residential structures, and their family members.

The study data will allow identifying (a) whether the social distancing between family members/caregivers and patients undergoing rehabilitation for orthopedic or neurological disabilities affects the quality of life and the emotional-affective sphere and (b) if these conditions change over time. The data obtained will, therefore, allow identifying those subjects who present a particular fragility of the emotional-affective sphere and who therefore need attention and possibly psychological support that will be prescribed.

Procedures:

Demographic (for patients and caregivers) and anamnestic (only for patients) data will be collected; moreover, disability will be assessed in patients using the modified Barthel index.

Three questionnaires will be administered to patients and caregivers:

* The Short Form (36) Health Survey (SF36), to evaluate the QoL;
* The Beck Anxiety Inventory (BAI), to evaluate the emotional state;
* The Beck Depression Inventory-II (BDI-II), to evaluate mood.

These questionnaires will be administered after one month of hospitalization (T0), and after one (T1) and two (T2) months after T0. Finally, at time T1 and T2 it will be registered if the patient is still hospitalized or discharged (and in the latter case the days between the discharge and the compilation of the questionnaire will be recorded). Since the three selected questionnaires provide for self-administration, to simplify the collection of data relating to caregivers, the implementation and use of an online questionnaire will be assessed. This questionnaire will also provide for the collection of consent to the use of data by the subject and will guarantee their privacy.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the centers of the Don Gnocchi Foundation participating in the study and their caregivers will be recruited

Exclusion Criteria:

* For patients: a score on the Mini-Mental State Examination (MMSE) scale lower than 24 which prevents the administration of SF36;
* For patients and caregivers: failure to acquire informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to inpatients rehabilitation centers
  Caregivers of patients admitted to inpatients rehabilitation centers
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Short Form-36 Health Survey (SF36) | After one month of hospitalisation (baseline, T0)
  It is a questionnaire to evaluate the Quality of Life
Short Form (36) Health Survey (SF36) | One month after baseline (T1)
  It is a questionnaire to evaluate the Quality of Life
Short Form (36) Health Survey (SF36) | Two months after baseline (T2)
  It is a questionnaire to evaluate the Quality of Life
Beck Anxiety Inventory (BAI) | After one month of hospitalisation (baseline,T0)
  It is a brief, criteria-referenced assessment for measuring anxiety severity and level
Beck Anxiety Inventory (BAI) | One month after baseline (T1)
  It is a brief, criteria-referenced assessment for measuring anxiety severity and level
Beck Anxiety Inventory (BAI) | Two months after baseline (T2)
  It is a brief, criteria-referenced assessment for measuring anxiety severity and level
Beck Depression Inventory-II (BDI-II) | After one month of hospitalisation (baseline)
  It is a brief, criteria-referenced assessment for measuring depression severity
Beck Depression Inventory-II (BDI-II) | One month after baseline (T1)
  It is a brief, criteria-referenced assessment for measuring depression severity
Beck Depression Inventory-II (BDI-II) | Two months after baseline (T2)
  It is a brief, criteria-referenced assessment for measuring depression severity

SECONDARY OUTCOMES:
modified Barthel Index (mBI) | After one month of hospitalisation (baseline, T0)
  It is a measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Irene APRILE, MD,PHD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Don Gnocchi Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Aprile I, Piazzini DB, Bertolini C, Caliandro P, Pazzaglia C, Tonali P, Padua L. Predictive variables on disability and quality of life in stroke outpatients undergoing rehabilitation. Neurol Sci. 2006 Apr;27(1):40-6. doi: 10.1007/s10072-006-0563-5. PMID 16688598